CLINICAL TRIAL: NCT06570876
Title: Radical Versus Conservative Surgery in Liver Cystic Echinococcosis: a Prospective Cohort Study in a High-volume Western Centre
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Marina Vila Tura, Marina Vila Tura, MD, Hospital Universitari de Bellvitge
Other Study IDs: PR048/23
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Liver; Cyst, Hydatid, Granulosus (Etiology)
Keywords: Liver cystic echinococcosis; Liver hydatid; Hepatic resection; Hepatic surgery; Biliary fistula; Bile leakage; Recurrence; Risk factor
MeSH Terms: conditions — Cysts; Biliary Fistula; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radical surgery: Total cystopericystectomy and anatomical liver resections are considered RS (i.e., segmentectomy, bisegmentectomy, left lateral segmentectomy, left hepatectomy, right hepatectomy, right trisectionectomy, and liver transplantation).
  Interventions: Procedure: Surgery
- Conservative surgery: Partial cystopericystectomy and the Lagrot technique are considered CS.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — The decision between RS and CS depended on the patient's performance status; on the cyst's main characteristics and contact with liver structures; and on intraoperative findings.

SUMMARY:
The goal of this observational study is to compare the results in terms of morbidity and disease-free survival between groups of patients with liver cystic echinococcosis (LCE) managed with radical surgery (RS) or conservative surgery (CS), and to evaluate potential risk factors of clinically relevant biliary fistula and liver recurrence.

DETAILED DESCRIPTION:
Main hypothesis:

1. Radical surgery (RS) in LCE has better postoperative results than conservative surgery (CS) in terms of global morbidity, specific morbidity and liver recurrence rate.

   Secondary hypotheses:
2. It is possible to identify preoperative and intraoperative prognostic factors of higher morbidity and recurrence rate.
3. The location of the residual pericystic layer in CS is related to a higher incidence of liver recurrence.
4. The percentage of residual pericystic layer in CS is related to a higher incidence of postoperative biliary fistula.

Main outcome:

1. To assess the incidence of liver recurrence between the RS and the CS groups, identifying potential risk factors.
2. To evaluate the incidence of postoperative biliary fistula between the RS and the CS groups, identifying possible risk factors.

Secondary outcomes:

1. To estimate the incidence of overall morbidity related to surgery.
2. To estimate the incidence of specific morbidity related to surgery (biliary fistula, intra-abdominal abscess, residual cavity abscess, hemoperitoneum, incisional infection, liver failure, respiratory infection, others).
3. To specifically analyze the incidence of postoperative biliary fistula and complex biliary fistula, and identify possible risk factors.
4. To estimate the incidence of mortality related to surgery.
5. To estimate the rate of hepatic and extrahepatic recurrence (number of disease-free months)
6. Prepare a recommendation for a standardized management algorithm for LCE patients based on the results obtained in the study and make it applicable to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult population (18 years or older) of both sexes surgically intervened for a diagnosis of LCE at the Bellvitge University Hospital and during the period described using a conservative or radical technique.
* Patients with asymptomatic liver hydatid cysts of active type or transition CE1 to CE3 according to the WHO classification.
* Patients with symptomatic or complicated hepatic hydatid cysts of any type (CE1 to CE5) according to the WHO classification.

Exclusion Criteria:

* Patients under 18 years of age.
* Patient operated on for LCE diagnosis with inactive asymptomatic cysts (CE4 or CE5 according to the WHO classification).
* Patients with less than 1 year of follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospective analysis of patients who undergo surgery for LCE from January 1996 to December 2021 at the Hepatobiliary Surgery and Liver Transplantation Unit of the Bellvitge University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 1996-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of liver recurrence between the RS and the CS groups, identifying potential risk factors | Diagnosis during the first 6 months was considered as persistence of the disease.
  Hepatic recurrence was defined as the appearance of a new growing cyst, non-detected by radiologic exploration before the first surgery, in the first location of the hydatid cyst in the liver or in another liver's segment.
To evaluate the incidence of postoperative biliary fistula between the RS and the CS groups, identifying possible risk factors. | 90 days postoperative
  The type of fistula was classified according to the International Study Group of Liver Surgery classification. A complex biliary fistula was defined as external bile leakage for ≥28 days and/or the need for percutaneous drainage or reoperation.

SECONDARY OUTCOMES:
To estimate the incidence of overall morbidity related to surgery. | 90 days postoperative
To estimate the incidence of specific morbidity related to surgery. | 90 days postoperative
  Biliary fistula, intra-abdominal abscess, residual cavity abscess, hemoperitoneum, incisional infection, liver failure, respiratory infection, others).
To specifically analyze the incidence of postoperative biliary fistula and complex biliary fistula, and identify possible risk factors. | 90 days postoperative
To estimate the incidence of mortality related to surgery. | 90 days postoperative
To estimate the rate of hepatic and extrahepatic recurrence (number of disease-free months) | From 6 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Marina Vila Tura, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McManus DP, Zhang W, Li J, Bartley PB. Echinococcosis. Lancet. 2003 Oct 18;362(9392):1295-304. doi: 10.1016/S0140-6736(03)14573-4. PMID 14575976
- [Background] Gollackner B, Langle F, Auer H, Maier A, Mittlbock M, Agstner I, Karner J, Langer F, Aspock H, Loidolt H, Rockenschaub S, Steininger R. Radical surgical therapy of abdominal cystic hydatid disease: factors of recurrence. World J Surg. 2000 Jun;24(6):717-21. doi: 10.1007/s002689910115. PMID 10773125
- [Background] Beyrouti MI, Beyrouti R, Bouassida M, Ben Amar M, Frikha F, Ben Salah K, Abid B, Guirat A, Ghorbel A, Mnif J, Ayadi A. [Hydatid cysts of the spigelian lobe (segment I) of the liver: clinical and therapeutic particularities]. Presse Med. 2007 Dec;36(12 Pt 1):1732-7. doi: 10.1016/j.lpm.2007.03.047. Epub 2007 Oct 31. French. PMID 17976950
- [Background] El Malki HO, El Mejdoubi Y, Souadka A, Mohsine R, Ifrine L, Abouqal R, Belkouchi A. Predictive factors of deep abdominal complications after operation for hydatid cyst of the liver: 15 years of experience with 672 patients. J Am Coll Surg. 2008 Apr;206(4):629-37. doi: 10.1016/j.jamcollsurg.2007.11.012. Epub 2008 Jan 28. PMID 18387467
- [Background] Wen H, Vuitton L, Tuxun T, Li J, Vuitton DA, Zhang W, McManus DP. Echinococcosis: Advances in the 21st Century. Clin Microbiol Rev. 2019 Feb 13;32(2):e00075-18. doi: 10.1128/CMR.00075-18. Print 2019 Mar 20. PMID 30760475
- [Background] Kratzer W, Weimer H, Schmidberger J. Echinococcosis: a Challenge for Liver Sonography. Ultraschall Med. 2022 Apr;43(2):120-145. doi: 10.1055/a-1694-5552. Epub 2022 Feb 24. PMID 35211944
- [Background] Farhat W, Ammar H, Rguez A, Harrabi F, Said MA, Ghabry L, Gupta R, Ben Cheikh A, Ghali H, Ben Rajeb M, Ben Mabrouk M, Ben Ali A. Radical versus conservative surgical treatment of liver hydatid cysts: A paired comparison analysis. Am J Surg. 2022 Jul;224(1 Pt A):190-195. doi: 10.1016/j.amjsurg.2021.12.014. Epub 2021 Dec 16. PMID 34949334
- [Background] Pang Q, Jin H, Man Z, Wang Y, Yang S, Li Z, Lu Y, Liu H, Zhou L. Radical versus conservative surgical treatment of liver hydatid cysts: a meta-analysis. Front Med. 2018 Jun;12(3):350-359. doi: 10.1007/s11684-017-0559-y. Epub 2017 Nov 23. PMID 29170917